CLINICAL TRIAL: NCT03132805
Title: An Evaluation of an Integrated Approach to Prevention and Early Intervention in the Elementary School Years
Acronym: P2P+IY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: DA039869; R01DA039869 (NIH)
Record Dates: First submitted 2017-04-04; First posted 2017-04-28 (Actual); Results first posted 2022-07-29 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Aggression
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: Schools are randomly assigned to 1 of 3 conditions, control, universal classroom-based preventive intervention, and universal classroom-based intervention plus an indicated preventive intervention. Data on student outcomes to be collected at pre- post- and 6 month follow-up. *Enrollment numbers reflect both students and teachers who agreed to participate in the study.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blind to intervention status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Schools which receive no intervention
- PATHS to PAX (Experimental): Universal classroom-based preventive intervention designed to reduce aggression.
  Interventions: Behavioral: PATHS to PAX
- PATHS to PAX and the IncredibleYears (Experimental): The combination of PATHS to PAX with the Incredible Years child and parent groups.
  Interventions: Behavioral: PATHS to PAX and the Incredible Years

INTERVENTIONS:
Behavioral: PATHS to PAX — A universal classroom-based preventive intervention designed to prevent aggression.
  Arms: PATHS to PAX
Behavioral: PATHS to PAX and the Incredible Years — A universal classroom-based preventive intervention in combination with an indicated preventive intervention, both of which are designed to prevent aggression.
  Arms: PATHS to PAX and the IncredibleYears

SUMMARY:
In this study, the investigators propose to examine whether the combination of a universal, elementary school-based preventive intervention with an indicated preventive and treatment intervention would yield greater impact on aggression than the universal preventive intervention alone.

DETAILED DESCRIPTION:
Aggressive behavior in the elementary school years is a strong indicator of antisocial behavior, drug abuse and low educational and occupational attainment in adolescence and young adulthood. The Good Behavior Game (GBG) and Promoting Alternative Thinking Strategies (PATHS) represent two of a handful of universal, elementary school, preventive interventions which have been shown in large scale, randomized controlled trials to have an immediate and beneficial impact on aggression. Promoting Alternative Thinking Strategies seeks to accomplish reductions in aggressive behavior via teacher led instruction aimed at facilitating emotion regulation and social problem-solving, whereas the Good Behavior Game provides teachers with an efficient means of reducing aggressive behavior using social learning principles within a game-like context. Importantly, however, the effects of the Good Behavior Game on aggressive behavior proved modest in the first and second generation Johns Hopkins University Preventive Intervention Research Center randomized field trials. This has been the case for Promoting Alternative Thinking Strategies as well. The investigators recently completed a 27-school, randomized controlled trial examining whether the combination of these interventions, which the investigators refer to as PATHS to PAX, would yield significantly greater impact on aggressive behavior than the Good Behavior Game alone. The rationale for expecting greater impact was that the use of the Good Behavior Game should result in reductions in aggressive behavior, which should then facilitate the acquisition of the emotion regulation and social problem-solving skills taught in Promoting Alternative Thinking Strategies. PATHS to PAX did result in a modestly greater reduction in aggressive behavior than the Good Behavior Game alone at 1-year post-test. Yet, the most aggressive students still failed to sufficiently benefit from the PATHS to PAX intervention. Accordingly, in this application, the investigators propose to examine whether the addition of the Incredible Years (IY), an evidence-based preventive and treatment intervention aimed at reducing aggressive behavior, to PATHS to PAX would yield greater impact on these behaviors than the PATHS to PAX intervention alone. The investigators also propose to examine whether the combination of the PATHS to PAX plus the Incredible Years results in increased frequency of implementation of the PATHS to PAX intervention. It is hypothesized that relative to teachers in the PATHS to PAX alone condition, teachers in the PATHS to PAX plus Incredible Years condition will perceive PATHS to PAX as more efficacious and will therefore be more likely to implement it. Four cohorts of 12 schools each will be recruited with schools randomly assigned to 1 of 3 intervention conditions: 1) Control; 2) PATHS to PAX; or 3) PATHS to PAX plus the Incredible Years. Assessments of student outcomes will be carried out at pre-test and post-test in the fall and spring of the initial school year for each cohort and at a 6-month and 1-year follow-up. Teacher outcomes in terms of classroom behavior management self-efficacy, perceptions of the efficacy of PATHS to PAX, and teacher burn out will be assessed at 4-time points during the initial year for each cohort. Assessment of teacher implementation of PATHS to PAX will be carried out on a daily basis throughout the intervention year. Aims 1 and 2 represent the primary goals of this application, whereas Aims 3 and 4 represent secondary, or exploratory, aims:

1. To evaluate, utilizing a group randomized design, whether the combination of PATHS to PAX plus Incredible Years child and parent groups yields greater reductions in aggressive behavior than PATHS to PAX alone.
2. To examine whether the frequency of PATHS to PAX intervention implementation (i.e., number of times and minutes the Good Behavior Game is played per day and Promoting Alternative Thinking Strategies lessons taught per week) will be greater in the PATHS to PAX plus Incredible Years condition.
3. To explore whether any evidence of differential benefits in terms of student outcomes between the PATHS to PAX versus PATHS to PAX plus Incredible Years conditions at post-test are a function of differences in PATHS to PAX implementation (e.g., number of Promoting Alternative Thinking Strategies lessons administered and the number of Good Behavior Games played and the duration of the games played). In addition, the investigators will explore whether any differences in implementation across the two intervention conditions is mediated by differences in teacher behavior management self-efficacy, perceived efficacy of PATHS to PAX in improving student behavior, and teacher burn out at post-test.
4. To explore the moderating effects of teacher, parent and student characteristics on intervention outcomes by expanding the models used for Aims 1 & 2 to include interactions between those characteristics and study condition,

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in kindergarten through second grade classrooms and their teachers.

Exclusion Criteria:

* Students must be enrolled in regular education classrooms.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5233 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Ialongo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1997). Maslach Burnout Inventory: Third edition. In C. P. Zalaquett & R. J. Wood (Eds.), Evaluating stress: A book of resources (pp. 191-218). Scarecrow Education.
- [Background] Tapp, J., Wehby, J., & Ellis, D. (1995). A multiple option observation system for experimental studies: MOOSES. Behavior Research Methods, Instruments & Computers, 27(1), 25-31.
- [Background] Harter S, Pike R. The pictorial scale of perceived competence and social acceptance for young children. Child Dev. 1984 Dec;55(6):1969-82. PMID 6525886
- [Background] Main, S., & Hammond, L. (2008). Best Practice or Most Practiced? Pre-Service Teachers' Beliefs about Effective Behaviour Management Strategies and Reported Self-Efficacy. Australian Journal of Teacher Education, 33, 28-39.
- [Background] Werthamer-Larsson L, Kellam S, Wheeler L. Effect of first-grade classroom environment on shy behavior, aggressive behavior, and concentration problems. Am J Community Psychol. 1991 Aug;19(4):585-602. doi: 10.1007/BF00937993. PMID 1755437
- [Background] Domitrovich CE, Bradshaw CP, Berg JK, Pas ET, Becker KD, Musci R, Embry DD, Ialongo N. How Do School-Based Prevention Programs Impact Teachers? Findings from a Randomized Trial of an Integrated Classroom Management and Social-Emotional Program. Prev Sci. 2016 Apr;17(3):325-37. doi: 10.1007/s11121-015-0618-z. PMID 26749578

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In accordance with our original protocol, we successfully recruited 48 schools over the four cohorts, which were subsequently randomized to one of three conditions. Randomization occurred at the school level and not at the teacher or student level within school. A total of 4,923 students with parental consent to participate were enrolled over the four cohorts from the 48 participating schools. A total of 310 teachers were also enrolled over the four cohorts from the 48 participating schools.
Units Other Than Participants: Schools
Period: Overall Study
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
Started (Students and teachers enrolled within participating schools) | 1629; 16 Schools | 1792; 16 Schools | 1812; 16 Schools
Students | 1527; 16 Schools | 1694; 16 Schools | 1702; 16 Schools
Teachers | 102; 16 Schools | 98; 16 Schools | 110; 16 Schools
Baseline Data Collection (Students) | 1442; 16 Schools | 1603; 16 Schools | 1617; 16 Schools
Post-test Data Collection (Students) | 1395; 16 Schools | 1564; 16 Schools | 1609; 16 Schools
Baseline Data Collection (Teachers) | 102; 16 Schools | 91; 16 Schools | 99; 16 Schools
Post-test Data Collection (Teachers) | 92; 16 Schools | 87; 16 Schools | 90; 16 Schools
Completed (Students and teachers enrolled within participating schools who were assessed at post-test) | 1487; 16 Schools | 1651; 16 Schools | 1699; 16 Schools
Not Completed | 142; 0 Schools | 141; 0 Schools | 113; 0 Schools
Not completed — Lost to Follow-up | 142 | 141 | 113

BASELINE CHARACTERISTICS:
Population: Students and teachers enrolled within participating schools who were assessed at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears | Total
Number analyzed (Participants) | 1544 | 1694 | 1716 | 4954
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline characteristics of enrolled students and enrolled teachers are represented on different rows.
  Participants
    Students: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    Students: <=18 years | 1442 | 1603 | 1617 | 4662
    Students: Between 18 and 65 years | 0 | 0 | 0 | 0
    Students: >=65 years | 0 | 0 | 0 | 0
    Teachers: number analyzed (Participants) | 102 | 91 | 99 | 292
    Teachers: <=18 years | 0 | 0 | 0 | 0
    Teachers: Between 18 and 65 years | 102 | 91 | 99 | 292
    Teachers: >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics of enrolled students and enrolled teachers are represented on different rows.
  Participants
    Students: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    Students: Female | 725 | 820 | 847 | 2392
    Students: Male | 717 | 783 | 770 | 2270
    Teachers: number analyzed (Participants) | 102 | 91 | 99 | 292
    Teachers: Female | 92 | 86 | 92 | 270
    Teachers: Male | 10 | 5 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics of enrolled students and enrolled teachers are represented on different rows.
  Participants
    Students: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    Students: Hispanic or Latino | 155 | 165 | 42 | 362
    Students: Not Hispanic or Latino | 1287 | 1438 | 1575 | 4300
    Students: Unknown or Not Reported | 0 | 0 | 0 | 0
    Teachers: number analyzed (Participants) | 102 | 91 | 99 | 292
    Teachers: Hispanic or Latino | 2 | 2 | 2 | 6
    Teachers: Not Hispanic or Latino | 100 | 89 | 97 | 286
    Teachers: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics of enrolled students and enrolled teachers are represented on different rows.
  Participants
    Students: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    Students: American Indian or Alaska Native | 7 | 25 | 10 | 42
    Students: Asian | 12 | 11 | 14 | 37
    Students: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Students: Black or African American | 1208 | 1341 | 1469 | 4018
    Students: White | 215 | 226 | 124 | 565
    Students: More than one race | 0 | 0 | 0 | 0
    Students: Unknown or Not Reported | 0 | 0 | 0 | 0
    Teachers: number analyzed (Participants) | 102 | 91 | 99 | 292
    Teachers: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Teachers: Asian | 3 | 4 | 1 | 8
    Teachers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Teachers: Black or African American | 58 | 41 | 47 | 146
    Teachers: White | 34 | 38 | 46 | 118
    Teachers: More than one race | 2 | 2 | 2 | 6
    Teachers: Unknown or Not Reported | 5 | 6 | 3 | 14
Region of Enrollment [Number; unit: Participants - Students & Teachers] — Population: Baseline characteristics of enrolled students and enrolled teachers are represented in the same row.
  Participants - Students & Teachers
    United States | 1544 | 1694 | 1716 | 4954
Teacher Observation of Child Adaptation- Revised (TOCA-R) [Mean (Standard Deviation); unit: units on a scale] — Student adaptation to classroom task demands are rated by teachers over the last 3 weeks on a 6-point frequency scale (1 = almost never to 6 = almost always). The domains include authority acceptance (α= 0.96; min=1; max=6) and readiness to learn (α= 0.97; min=1; max=6). Authority acceptance items include classroom rule compliance, & readiness to learn items reflect attentive classroom behaviors (e.g. stays on task). The mean of the teacher ratings across the items making up each of these subscales was used in the outcome analyses. Higher scores on both subscales reflect greater adaptation. Population: Students enrolled within participating schools who were assessed at baseline. Only students were included in this part of the data collection.
  units on a scale
    Readiness to Learn: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    Readiness to Learn | 4.115 (1.381) | 4.290 (1.336) | 4.193 (1.363) | 4.202 (1.361)
    Authority Acceptance: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    Authority Acceptance | 5.074 (1.104) | 5.300 (0.9506) | 5.217 (1.021) | 5.201 (1.028)
Independent Classroom Observations of Student Behavior [Mean (Standard Deviation); unit: percentage of intervals observed] — Classroom observations were completed by independent observers. The behaviors observed were on-task and physical aggression. Behaviors were observed in 10 second intervals and were recorded as present if they occurred at least once during a 10 second interval. The per interval on-task and physical aggression scores could range from 0-1, with 0 signifying the behavior was not observed and 1 signifying the behavior was observed. The on-task and physical aggression scores used in the analyses were the average score across all of the 10-second intervals the student was observed. Population: Students enrolled within participating schools who were assessed at baseline. Only students were included in this part of the data collection.
  percentage of intervals observed
    On-Task: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    On-Task | 0.4921 (0.2690) | 0.5172 (0.2476) | 0.5379 (0.2783) | 0.5166 (0.2657)
    Physical Aggression: number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    Physical Aggression | 0.0021 (0.0124) | 0.0015 (0.0096) | 0.0020 (0.0115) | 0.0019 (0.0112)
Peer Assessment Inventory [Mean (Standard Deviation); unit: percentage of nominations received] — Individual students were read aloud the names of the other students in the classroom. The student being interviewed was asked if they knew the named student. The student was then asked whether the peer nomination descriptors fit the named student (Do you like [student]?, Do you play with [student]?, and Is (s)he one of your best friends?). The student's summary score reflected the mean percentage of nominations received across the 3 items (α=0.91). A higher percentage reflects a student received a greater number of nominations from classmates. Population: Students enrolled within participating schools who were assessed at baseline. Only students were included in this part of the data collection.
  percentage of nominations received
    number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    (all) | 0.812 (0.187) | 0.816 (0.173) | 0.816 (0.170) | 0.815 (0.177)
The Pictorial Scale of Perceived Competence and Acceptance For Young Children [Mean (Standard Deviation); unit: units on a scale] — Items on this instrument present two pictorial alternatives, one of a child displaying high competence in the social acceptance domain and one that depicts less competence. Students were asked which pictorial plate was most like him/her. After making that decision, the student is then asked if the chosen picture is "really true for me" and "sort of true for me." Each item is scored on a 4-point scale, 4 would be the most competent and 1 would designate the least competent. The mean of the items was used in the outcome analyses. The coefficient alpha for the mean score was 0.71. Population: Students enrolled within participating schools who were assessed at baseline. Only students were included in this part of the data collection.
  units on a scale
    number analyzed (Participants) | 1442 | 1603 | 1617 | 4662
    (all) | 3.352 (0.591) | 3.305 (0.614) | 3.328 (0.591) | 3.328 (0.599)
The Behavior Management Self-Efficacy Scale & The Social-Emotional Learning Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — The Behavior Management Self-Efficacy Scale (Main and Hammond 2008) included 14 items regarding classroom behavior management (e.g., I can manage a class very well; α= 0.918; min=1; max=5). The Social-Emotional Learning Efficacy Scale (Domitrovich, et al., 2016) included 8 items which focused on teachers' perceived efficacy to promote social-emotional skills in students (e.g., I am able to teach children to show empathy; α= 0.909; min=1; max=5). For each scale, item responses were provided on a 5-point Likert-type scale, & were averaged, higher scores indicating greater efficacy. Population: Teachers enrolled in within participating schools who were assessed at baseline. Only teachers were included in this part of the data collection.
  units on a scale
    Behavior Management Self-Efficacy Scale: number analyzed (Participants) | 102 | 91 | 99 | 292
    Behavior Management Self-Efficacy Scale | 3.80 (0.54) | 3.89 (0.55) | 3.83 (0.57) | 3.84 (0.55)
    Social-Emotional Learning Efficacy Scale: number analyzed (Participants) | 102 | 91 | 99 | 292
    Social-Emotional Learning Efficacy Scale | 3.57 (0.62) | 3.76 (0.53) | 3.65 (0.59) | 3.66 (0.59)
The Maslach Burnout Inventory [Mean (Standard Deviation); unit: units on a scale] — Teachers completed the Maslach Burnout Inventory (MBI;Maslach et al. 1997). One scale was used in the analyses: emotional exhaustion (9 items, e.g., I feel used up at the end of the workday, α=0.937; min=1; max=7). Responses were rated on a 7-point scale from never to every day and to create scale scores such that higher scores indicated greater emotional exhaustion (i.e., greater burnout). Therefore, low scores on emotional exhaustion were desired. Population: Teachers enrolled within participating schools who were assessed at baseline. Only teachers were included in this part of the data collection.
  units on a scale
    number analyzed (Participants) | 102 | 91 | 99 | 292
    (all) | 3.64 (1.58) | 3.62 (1.49) | 3.90 (1.47) | 3.72 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Change in Direct Classroom Observations of Student Behavior Between Pre-test and Post-test, 6 Months After the Pre-test.
Description: Classroom observations of student behavior were carried out by independent observers on two occasions, one week apart, at pre- and post-test respectively. The behaviors observed were on-task and physical aggression. Behaviors were observed in 10 second intervals and were recorded as present if they occurred at least once during a 10 second interval. The per interval on-task and physical aggression scores could range from 0-1, with 0 signifying the behavior was not observed and 1 signifying the behavior was observed. The on-task and physical aggression scores used in the analyses were the average score across all of the 10-second intervals the student was observed. (Adapted from Tapp, Wehby & Ellis, 1995).
Time Frame: The observations are carried out at pre-test and at post-test, 6 months after the pre-test.
Population: Students enrolled within participating schools with parental consent to participate in the trial who were observed at baseline and at post-test.
Measure: Mean (Standard Error); unit: percentage of intervals observed
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
Number analyzed (Participants) | 763 | 891 | 1129
percentage of intervals observed
  On-Task | 0.42 (0.03) | 0.446 (0.02) | 0.453 (0.02)
  Physical Aggression | 0.004 (0.001) | 0.001 (0.001) | 0.001 (0.001)

2. Primary Outcome: Teacher Ratings of Student On-task and Aggressive-disruptive Behavior in the Classroom.
Description: Change in Teacher Observation of Classroom Adaptation between pre-test and post-test, 6 months after the pre-test. Student adaptation to classroom task demands are rated by teachers over the last 3 weeks on a 6-point frequency scale (1 = almost never to 6 = almost always). The domains include authority acceptance and readiness to learn. Authority acceptance items include compliance with classroom rules, and readiness to learn items reflect attentive classroom behaviors (e.g. stays on task). The mean of the teacher ratings across the items making up each of these subscales was used in the outcome analyses. The minimum score for both the authority acceptance and readiness to learn subscales was 1 and maximum score was 6. Higher scores on both subscales reflect greater adaptation.
Time Frame: The ratings are carried out at pre-test, post-test, 6 months after the pre-test.
Population: Students enrolled in participating schools with parental consent to participate in the trial who were teacher rated at baseline and post-test.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
Number analyzed (Participants) | 1316 | 1474 | 1531
score on a scale
  Readiness to Learn | 4.18 (0.09) | 4.50 (0.06) | 4.53 (0.09)
  Authority Acceptance | 4.98 (0.06) | 5.19 (0.07) | 5.14 (0.06)

3. Secondary Outcome: Change in Peer Assessment Inventory Between Pre-test and Post-test, 6 Months After the Pre-test.
Description: Students are asked to nominate fellow students in terms of who they like, play with, and perceive as friends. Individual students were read aloud the names of the other students in the classroom. The student being interviewed was asked if they knew the named student. The student was then asked whether the peer nomination descriptors fit the named student (Do you like [student]?, Do you play with [student]?, and Is (s)he one of your best friends?). The student's summary score reflected the mean percentage of nominations received across the 3 items. A higher percentage reflects a student received a greater number of nominations from classmates.
Time Frame: The peer nomination instrument is administered at pre-test and at post-test, 6 months after the pre-test.
Population: Students enrolled within participating schools with parental consent to participate in the trial who were interviewed at baseline and at post-test.
Measure: Mean (Standard Error); unit: percentage of nominations received
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
Number analyzed (Participants) | 847 | 918 | 1065
percentage of nominations received | 0.819 (0.02) | 0.806 (0.01) | 0.816 (0.02)

4. Secondary Outcome: Change in Pictorial Scale of Perceived Competence and Social Acceptance for Young Children Between Pre-test and Post-test, 6 Months After the Pre-test.
Description: The Change in Pictorial Scale of Perceived Competence and Social Acceptance for Young Children assesses the student's perceived competence in the domains of peer acceptance. Items on this instrument present two pictorial alternatives, one of a child displaying high competence in the social acceptance domain and one that depicts less competence. Students were asked which pictorial plate was most like him/her. After making that decision, the student is then asked if the chosen picture is "really true for me" and "sort of true for me." Each item is scored on a 4-point scale, 4 would be the most competent and 1 would designate the least competent. The mean of the items was used in the outcome analyses.
Time Frame: This scale will be administered at pre-test and post-test, 6-months after the pre-test.
Population: Students enrolled in participating schools with parental consent to participate in the trial who were interviewed at baseline and post-test.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
Number analyzed (Participants) | 847 | 918 | 1065
score on a scale | 3.36 (0.04) | 3.36 (0.03) | 3.41 (0.04)

5. Secondary Outcome: Change in Teacher Sense of Self Efficacy Scale Between Pre-test and Post-test, 6-months After the Pre-test.
Description: This scale assesses teacher sense of self-efficacy in the instructional and classroom behavior management domains. We assessed two distinct dimensions of teachers' perceived self-efficacy that reflect skills uniquely associated with the strategies included in the two interventions. The Behavior Management Self-Efficacy Scale (Main and Hammond 2008) included 14 items regarding classroom behavior management (e.g., I am able to use a variety of behavior management techniques; α= 0.92). The Social-Emotional Learning Efficacy Scale (Domitrovich, et al., 2016) included 8 items which focused on teachers' perceived efficacy to promote social-emotional skills in students (e.g., I am able to teach children to show empathy and compassion for each other; α= 0.91). For each scale, item responses were on a 5-point Likert-type scale and were averaged. For both subscales the minimum score was 1 and maximum was 5, with higher scores indicating greater efficacy.
Time Frame: This scale will be administered at pre-test and post-test, 6 months after the pre-test.
Population: Consenting teachers assigned to Kindergarten - second grade in participating trial schools who were assessed at baseline and post-test.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
Number analyzed (Participants) | 91 | 87 | 90
score on a scale
  Teacher Sense of Social Emotional Learning Self Efficacy | 3.56 (0.08) | 4.08 (0.09) | 3.92 (0.08)
  Teacher Sense of Behavior Management Self Efficacy | 3.82 (0.07) | 4.23 (0.07) | 4.09 (0.07)

6. Secondary Outcome: Change in the Maslach Burnout Inventory Between Pre-test and Post-test, 6 Months After the Pre-test.
Description: The Maslach Burnout Inventory assesses how frequently teachers experience feelings of burnout in the work place. Teachers completed the Maslach Burnout Inventory (MBI;Maslach et al. 1997) at pretest and post-test. One scale was used in the analyses: emotional exhaustion (9 items, e.g., I feel used up at the end of the workday, α=0.94). Responses were rated on a 7-point scale from never to every day with higher scores indicating greater emotional exhaustion (i.e., greater burnout). For this subscale, the minimum score was 1 and maximum score was 7. Therefore, low scores on emotional exhaustion were desired.
Time Frame: This scale will be administered at pre-test and post-test, 6 months after the pre-test.
Population: as for outcome 5
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
Number analyzed (Participants) | 91 | 87 | 90
score on a scale | 4.02 (0.19) | 3.10 (0.23) | 3.40 (0.20)

ADVERSE EVENTS:
Time Frame: Over the four year intervention implementation phase of the trial.
Description: No difference
Arm/Group | Control | PATHS to PAX | PATHS to PAX and the IncredibleYears
All-Cause Mortality (participants affected / at risk) | 0/1629 | 0/1792 | 0/1812
Serious Adverse Events (participants affected / at risk) | 0/1629 | 0/1792 | 0/1812
Other Adverse Events (participants affected / at risk) | 0/1629 | 0/1792 | 0/1812

LIMITATIONS AND CAVEATS:
Due to the COVID-19 school related disruptions, we were unable to fully complete the implementation of the interventions for the 4th cohort. We were unable to complete the Classroom Observations of Student Behavior, Peer Assessments, and Perceived Competence of Social Acceptance at post-test in the 4th cohort. The Teacher Observation of Classroom Adaptation scales were completed based on the virtual-learning environment for the one-year follow-up of the 4th cohort of students.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/05/NCT03132805/Prot_SAP_000.pdf